CLINICAL TRIAL: NCT00185744
Title: Accelerated Partial Breast Irradiation Following Lumpectomy for Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13807
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Carcinoma, Ductal
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal | interventions — Mastectomy, Segmental; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Accelerated Partial Breast Irradiation (Experimental): lumpectomy with accelerated partial breast irradiation
  Interventions: Radiation: Intra-Operative Radiotherapy (IORT); Procedure: Lumpectomy; Radiation: Intracavitary Brachytherapy; Radiation: Accelerated External Beam 3-D Conformal Radiotherapy; Radiation: Stereotactic APBI
- Standard Therapy (Active Comparator): lumpectomy and whole breast irradiation
  Interventions: Procedure: Lumpectomy; Radiation: Whole Breast Radiotherapy

INTERVENTIONS:
Radiation: Intra-Operative Radiotherapy (IORT) — single dose in the operating room after lumpectomy
  Arms: Accelerated Partial Breast Irradiation
Procedure: Lumpectomy
Radiation: Whole Breast Radiotherapy — six and a half week treatment
  Arms: Standard Therapy
Radiation: Intracavitary Brachytherapy — 5 day treatment
  Other Names: MammoSite
  Arms: Accelerated Partial Breast Irradiation
Radiation: Accelerated External Beam 3-D Conformal Radiotherapy — 5 day treatment
  Arms: Accelerated Partial Breast Irradiation
Radiation: Stereotactic APBI — 4 day treatment
  Arms: Accelerated Partial Breast Irradiation

SUMMARY:
To determine whether an accelerated course of radiotherapy delivered to the lumpectomy cavity plus margin using IORT as a single dose, intracavitary brachytherapy with the MammoSite device over 5 days, partial breast 3-D CRT in 5 days, or stereotactic APBI over 4 days is a feasible and safe alternative to a six and a half week course of whole breast radiotherapy. The study will measure both short and long-term complications of radiation treatment, short and long-term breast cosmesis, local rates of in-breast cancer recurrence, regional recurrences, distant metastases, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Women >= 40 with invasive ductal carcinoma or ductal carcinoma in situ
2. Patient chooses lumpectomy rather than mastectomy as treatment for breast cancer
3. Tumor < 2.5 cm in size, 2 mm margin of normal breast tissue between cancer and edge of specimen.

Exclusion Criteria:

1. Men
2. Prior malignancy, breast or other if metastatic or with anticipated survival of < 5 years
3. Pregnant women
4. Immunocompromised
5. Poorly controlled insulin dependent diabetes
6. Contraindication to radiotherapy, e.g. connective tissue disorder such as scleroderma
7. Breast cancer that involves skin or chest wall
8. Multifocal or Multicentric breast cancer
9. Invasive lobular carcinoma
10. Diffuse microcalcifications on mammography
11. Invasive carcinoma with extensive intraductal component (EIC)
12. Greater than 12 weeks since definitive surgical excision or completion of chemotherapy
13. Involved lymph nodes detected by frozen section or touch preparation at time of lumpectomy
14. Patients with 1 to 3 positive lymph nodes determined postoperatively (does not include patients with micro-metastases)
15. Subglandular or submuscular breast implants (does not include patients having implants placed AFTER intra-operative radiotherapy)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-09; Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
In-breast tumor recurrence (IBTR) | 20 years
  Proportion of subjects that experience in-breast tumor recurrence (IBTR), to be assessed through or by March 2029

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M. Dirbas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horst KC, Fasola C, Ikeda D, Daniel B, Ognibene G, Goffinet DR, Dirbas FM. Five-year results of a prospective clinical trial investigating accelerated partial breast irradiation using 3D conformal radiotherapy after lumpectomy for early stage breast cancer. Breast. 2016 Aug;28:178-83. doi: 10.1016/j.breast.2016.06.001. Epub 2016 Jun 17. PMID 27322859